CLINICAL TRIAL: NCT05031403
Title: Development and Application of Tele-Neuro Rehabilitation System: An Example of Digital Transformation in Health
Brief Title: Development and Application of Tele-Neuro Rehabilitation System
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Istanbul University - Cerrahpasa (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, Yonca Zenginler Yazgan, Principal Investigator, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 120S843
Record Dates: First submitted 2021-07-05; First posted 2021-09-01 (Actual); Last update posted 2021-09-01 (Actual); Status verified 2021-07

CONDITIONS: Stroke; Multiple Sclerosis; Parkinson Disease
Keywords: E-Health; Web Based Systems; Neurologic Rehabilitation; Neurorehabilitation; Physical Therapy and Rehabilitation; Stroke Rehabilitation; Multiple Sclerosis; Parkinson's Disease; Data Storage; Stroke
MeSH Terms: conditions — Stroke; Multiple Sclerosis; Parkinson Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Stroke (Telerehabilitation) (Experimental): Exercise therapy with telerehabilitation system
  Interventions: Other: Telerehabilitaton
- Stroke (Home Exercise) (Other): Exercise therapy with brochure
  Interventions: Other: Home Exercise
- Multiple Sclerosis (Telerehabilitation) (Experimental): Exercise therapy with telerehabilitation system
  Interventions: Other: Telerehabilitaton
- Multiple Sclerosis (Home Exercise) (Other): Exercise therapy with brochure
  Interventions: Other: Home Exercise
- Parkinson Disease (Telerehabilitation) (Experimental): Exercise therapy with telerehabilitation system
  Interventions: Other: Telerehabilitaton
- Parkinson Disease (Home Exercise) (Other): Exercise therapy with brochure
  Interventions: Other: Home Exercise

INTERVENTIONS:
Other: Telerehabilitaton — Patients will be asked to apply the rehabilitation program defined for them 3 days a week for 8 weeks. A training session will last approximately 45-60 minutes.
  Arms: Multiple Sclerosis (Telerehabilitation); Parkinson Disease (Telerehabilitation); Stroke (Telerehabilitation)
Other: Home Exercise — Patients will be asked to apply the rehabilitation program for themselves with an exercise brochure. This therapy will last 3 days a week for 8 weeks.
  Arms: Multiple Sclerosis (Home Exercise); Parkinson Disease (Home Exercise); Stroke (Home Exercise)

SUMMARY:
Disability due to neurological diseases is increasing in our country and world. With regular physiotherapy and rehabilitation, as well as patients' symptoms are brought under control, their affected functions in daily life are achieved and levels of independence and physical activity increase. Thus, the patients' quality of life and participation in social life is improved and patients are supported in physical, social and psychological terms. In recent years, it has been reported that exercise with telerehabilitation systems increase the compliance and participation of patients to the treatment, and even this system seems as effective as standard rehabilitation practices. Delivering the treatment through telerehabilitation system when that patients cannot receive it in the hospital due to epidemic, restriction, transfer difficulties, personal and environmental limitations will enable patients to receive the rehabilitation services.Telerehabilitation system is frequently encountered in the abroad, but there are limited systems with Turkish version specific to this patient group in our country. The aim of project is to develop and detect the efficiency of a telerehabilitation system which is used to assess, follow and design home-based rehabilitation program among individuals with chronic neurological diseases who have difficulty in participating in physiotherapy and rehabilitation services because of personal or environmental reasons.

DETAILED DESCRIPTION:
The coding and design of this telerehabilitation system will enable easy access to all devices via the website. The expert interface of the system will consist of three interfaces; exercise videos to be prepared by physiotherapists will be uploaded, patient list and feedback of patients. Rehabilitation programs can be prepared and updated. There will be a panel in the patient interface that will allow the patient to access a rehabilitation program tailored to the problem and to communicate about the ongoing program when needed. In the manager interface, high-level control of many steps such as adding experts from different institutions, organizing information, creating an exercise pool will be provided. With the project, a telerehabilitation system will be put into practice, where patients can easily access the rehabilitation services from their homes, and patients can contact with clinicians when they need follow-up and treatment.

The patients and their caregivers will be informed about the system and project. In the assessment part, the physical performance will be determined. Also, questionnaires such as fall efficacy or activities of daily living will be requested through the system. Thus, a detailed assessment of the patient will be completed to reveal the problems. A rehabilitation program with appropriate exercises will be defined for patients in the telerehabilitation group and patients will be asked to apply this program three days a week for eight weeks. Patients in the control group will be placed on the waiting list after the first evaluations and no additional treatment will be applied by asking them to maintain their routine activity levels within this period. At the end of eight weeks, initial evaluations will be repeated in two groups.

This user-friendly telerehabilitation system with turkish language support will be the first comprehensive system that will let to assess, give exercise programs and follow the progression in patients with chronic neurologic disorders. With this system, the opportunity to reach more patients in the home environment will be provided. Rehabilitation programs will promote the physical capacity, health-related quality of life and it will also cause reducing in the burden of caregivers. After evaluating the applicability of our program, we will pave the way for the introduction of telerehabilitation care in health institutions and in areas with transportation issues, furthermore low-cost, sustainable system will be achieved to our country.

ELIGIBILITY:
Inclusion Criteria:

* Chronic patients diagnosed with neurological disease at least 1 year ago by a neurologist
* Multiple sclerosis patients with an Expanded Disability Status Scale (EDSS) score of ≤6, who are in the stable phase of the disease and have not had an attack in the last 3 months
* Parkinson's patients with a Hoehn and Yahr score ≤3
* Stroke patients with a modified Rankin score of ≤3
* To have an internet infrastructure where the system can be accessed at home
* Not participating in a standardized physiotherapy and rehabilitation program within the last 3 months
* Having a companion with the patient during the exercises

Exclusion Criteria:

* Presence of blurred or poor vision problems
* Hearing and speech impairment at a level that will affect participation in the system
* Epilepsy
* The presence of pregnancy
* Having any cognitive problems that prevent using the system
* History of trauma / fracture in the last 3-6 months
* Having pacemaker
* Presence of cardiac problems
* Presence of serious respiratory diseases

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-09-01 (Estimated); Study Completion 2022-10-01 (Estimated)

PRIMARY OUTCOMES:
Independent Standing Test (The change between the initial value and the value after 2 months will be evaluated). | Baseline and end of weeks 8.
  It tests the patient's ability to stand for 20 seconds in an upright position without any support or assistance, with her/his feet shoulder-width apart and arms free at the side of the body.
Romberg Test (The change between the initial value and the value after 2 months will be evaluated). | Baseline and end of weeks 8.
  The patient is asked to stand in an upright position with his feet open at shoulder level, arms free at the side of the body, with eyes open and then closed, without losing his balance for 10 seconds before receiving any support. In case of excessive release or failure to continue the test, it is considered a Romberg positive or abnormal Romberg sign. It evaluates the effect of the patient's balance in the closed position.
One-Legged Standing Test (The change between the initial value and the value after 2 months will be evaluated). | Baseline and end of weeks 8.
  It is a functional evaluation test that measures the patient's one-leg standing balance. The patient is asked to raise one leg in the air and keep the knee bent at hip level for at least 10 seconds. Times less than 10 seconds indicate a balance disorder, and times less than 5 seconds indicate a risk of falling. It is applied with the patient's eyes open and closed.
5 Times Sit and Stand Test (The change between the initial value and the value after 2 months will be evaluated). | Baseline and end of weeks 8.
  It is a test that evaluates functional lower extremity strength, transfer, balance and fall risk. The time for the patient to sit and stand up from the chair 5 times is recorded. It has been proven to be valid in patients with stroke, Parkinson's and Multiple Sclerosis.
KATZ Independence Index in Activities of Daily Living (The change between the initial value and the value after 2 months will be evaluated). | Baseline and end of weeks 8.
  It is a scale that measures the ability of the patient to do daily living activities independently and evaluates the functional status. It examines patient performances in six functions such as bathing, dressing, toilet, transfer, personal care and feeding. Patients score their activity independence in each of the six functions as 1 (independent) or 0 (dependent). A total score of 0 to 2 indicates severe dysfunction, a total score of 2 to 4 indicates moderate dysfunction, and a total score of 4 to 6 indicates full function.

SECONDARY OUTCOMES:
Modified Fall Efficiency Scale (The change between the initial value and the value after 2 months will be evaluated). | Baseline and end of weeks 8.
  It is a 14-item scale that measures the patient's confidence in falling. Each question is scored between 1-4. High scores indicate high fall anxiety.
World Health Organization Quality of Life Scale Short Form Turkish Version (WHOQOL-BREF-TR) (The change between the initial value and the value after 2 months will be evaluated). | Baseline and end of weeks 8.
  It is a health-related quality of life scale developed by the World Health Organization. A national question was added to the Turkish version of the scale in addition to the original version. The scale measures physical, mental, social and environmental well-being and consists of a total of 27 questions with an additional question. Since each domain independently expresses the quality of life in its own field, field scores are calculated between 4-20. The higher the total score, the higher the quality of life.
Fatigue Severity Scale (The change between the initial value and the value after 2 months will be evaluated). | Baseline and end of weeks 8.
  It is a scale that evaluates the severity of fatigue with 9 items that patients can answer on their own. Each item is scored between 1 (strongly disagree) and 7 (strongly agree). The total score is calculated by taking the average of 9 items. A high score indicates increased fatigue severity.
System Usability Scale (The change between the initial value and the value after 2 months will be evaluated). | Baseline and end of weeks 8.
  It is a scale consisting of 10 questions widely used in the literature to evaluate the perceptibility and usability of interactive systems. It is scored from 1 (strongly disagree) to 5 (strongly agree). A high total score indicates that the system is detectable and usable.
Global Change Scale (The change between the initial value and the value after 2 months will be evaluated). | Baseline and end of weeks 8.
  It is a scale that evaluates how much a person's current situation has changed compared to his previous state. The person is asked to choose an exchange score from -5 (much worse than my previous state) to +5 (much better than my previous state).

CONTACTS AND LOCATIONS:
Overall Officials: Ela Tarakcı, Prof., Study Chair — Istanbul University-Cerrahpaşa Faculty of Health Sciences; Burcu Ersöz Hüseyinsinoğlu, Assoc. Prof, Study Chair — Istanbul University-Cerrahpaşa Faculty of Health Sciences; Murat Kürtüncü, MD, Study Chair — Istanbul University-Capa Faculty of Medicine, Department of Neurology; Muhammed Erdem İsenkul, Asst. Prof., Study Chair — Istanbul University-Cerrahpaşa Faculty of Engineering; Pelin Vural, Study Chair — Istanbul University-Cerrahpasa Institute of Postgraduate Education; Recep Örmen, Study Chair — Istanbul University-Cerrahpasa Institute of Postgraduate Education
Locations (1):
- Istanbul University-Cerrahpasa, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No